CLINICAL TRIAL: NCT06631040
Title: Cell Therapy with Anti-CD19 CAR-NK Cells in Patients with Relapsed or Resistant B-Acute Lymphocytic Leukemia
Brief Title: Cell Therapy with Anti-CD19 CAR-NK Cells in Patients with Relapsed or Resistant B-ALL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Soleimani, Professor, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 75358
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Acute Lymphocytic Leukemia in Relapse
Keywords: CAR-NK Therapy; anti-CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute lymphocytic leukemia, in relapse (Experimental)
  Interventions: Biological: anti CD19 CAR NK cells

INTERVENTIONS:
Biological: anti CD19 CAR NK cells — Ten eligible patients with relapsed Acute Lymphoblastic Leukemia will be enrolled based on inclusion criteria and informed consent. After conditioning with Fludarabine and Cyclophosphamide, patients will receive a single infusion of anti-CD19 CAR NK cells with close monitoring using one of the following dose levels: • Dose Level 1: 1×10^7/Kg • Dose Level 2: 5×10^7/Kg • Dose Level 3: 1×10^8/Kg Safety Assessment: Adverse events will be recorded and graded. Laboratory parameters and cytokine release syndrome (CRS) markers will be closely monitored. Efficacy Evaluation: Response assessments will follow International Lymphoma Party (LWP) Group guidelines, including complete response (CR), partial response (PR), stable disease (SD), and progressive disease.

SUMMARY:
Immunotherapy has shown promise in treating hematological malignancies, including resistant B-ALL. One approach is CAR-NK cell therapy, which involves genetically modifying natural killer (NK) cells to target specific cancer antigens. While CAR-NK therapy offers advantages over CAR-T therapy, such as reduced immune system reactions and lower production time and cost, challenges remain regarding antitumor efficacy and the tumor microenvironment. Preclinical and early clinical studies have targeted various antigens, including CD19, with CAR-NK cells in resistant B-ALL. To further investigate the potential of anti-CD19 CAR-NK cell therapy, this study aims to evaluate its safety and determine the maximum tolerated dose (MTD) in patients who have not responded to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

Eligible diseases: Acute lymphocytic leukemia (ALL CD19+). Patients 3 years of age or older, and must have a life expectancy > 12 weeks. Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.

Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR NK cells.

Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.

Ability to give informed consent.

Exclusion Criteria:

Pregnant or nursing women may not participate. Active HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at the time of screening.

Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.

History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.

Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.

The existence of unstable or active ulcers or gastrointestinal bleeding. Patients need anticoagulant therapy (such as warfarin or heparin). Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).

Patients using fludarabine or cladribine chemotherapy within 3 months prior to leukapheresis.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-19 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLTs) | 4 weeks
  Incidence of dose-limiting toxicity (DLTs) within 4 weeks after infusion, characterized by >= Grade 3 signs/symptoms according to CTCAE v4.03, to assess safety and tolerability.
Assessment of Maximum Tolerated Dose (MTD) | 4 weeks
Overall Remission Rate (ORR) | 8 weeks
  Overall Remission Rate (ORR) two months after infusion, assessed using International lymphoma party (LWP) Group

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 48 weeks
  Assessed using International Lymphoma Working Party (LWP) criteria
Duration of Response (DOR) | 48 weeks
  Duration of Response (DOR) for up to 12 months, Assessed using International Lymphoma Working Party (LWP) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Ghazi Hospital, Tabriz university of medical sciences, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: Undecided